CLINICAL TRIAL: NCT00489892
Title: Efficacy of Pharmacological Treatment of Working Memory Impairment After Traumatic Brain Injury: Evaluation With fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: University of Medicine and Dentistry of New Jersey (Other); Cephalon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-437-02; 0120020166; M-166-2002
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Traumatic Brain Injury; Severe Traumatic Brain Injury
Keywords: traumatic brain injury; TBI; working memory; modafinil; fMRI; MRI
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
This study is designed to examine the effects of a wake-promoting agent (Modafinil) on working memory (WM) in persons with moderate to severe TBI utilizing a double blinded placebo controlled methodology. Our approach is to evaluate participants with BOLD fMRI and a limited neuropsychological battery to examine WM performance before and after pharmacological intervention.

Hypotheses

1. Because increased cognitive effort (as a function of decreased efficiency after TBI) is presumed to underlie fMRI activation dispersion that is seen during central executive WM tasks, we anticipate an attenuation of cerebral activation in prefrontal cortex during pharmacological intervention with Modafinil when compared to placebo administration on the mPASAT and vigilance testing.
2. There will be a correlation between the decreased dispersion of the fMRI signal on scans and improvement in neuropsychological measures when individuals are on Modafinil that is not seen when they are taking placebo.

DETAILED DESCRIPTION:
Work from our institution has shown that moderate and severe TBI subjects demonstrate an altered cerebral representation when they attempt to process a verbal WM task. Specifically, our data show a post-TBI pattern of activation that is dispersed and more lateralized to the right hemisphere, as compared to healthy controls. Taken together, we interpret these findings to mean that it is requires more cerebral resources for TBI subjects to process tasks that were previously more automatic. In other words, their processing is less efficient. This is consistent with TBI patients' self-reports of needing to expend greater cognitive effort to perform such tasks, both in the lab and in everyday life. Our preliminary data was the first step in understanding the cerebral substrate of these difficulties. However, simply indicating that individuals with TBI have a WM problem is not enough. The development of targeted interventions to ameliorate these deficits is the next step in the treatment process.

The present proposal has important implications for TBI rehabilitation. One of the major goals of cognitive remediation is to help TBI patients learn new information more accurately and efficiently, and to improve their performance in activities of everyday life. 123 Because WM impairments are so prevalent in TBI, the present study can help to shed light on potential treatment alternatives for these potentially devastating problems. In spite of the prevalence and popularity of cognitive remediation strategies and procedures, there remains little empirical support for their efficacy, and virtually no understanding of the underlying neurocognitive processes that facilitate intervention. The ability to develop a potentially efficacious treatment modality, which has a solid foundation, would be immensely beneficial.

ELIGIBILITY:
Inclusion Criteria:

We will include only those subjects who have sustained moderate to severe initial injuries, as defined by an initial 24-hour Glasgow Coma Scale 128 scores below 13. In the event that a GCS score is not available, subjects will only be included if there is sufficient medical documentation that would allow for a post-hoc estimation of initial GCS, or if other confirmatory data (e.g., positive anatomic neuroimaging findings, focal neurologic signs) are available. Individuals with a history of prior moderate to severe head injury, stroke, seizures, severe psychiatric disturbances (i.e., those known to influence memory performance, such as schizophrenia, bipolar disorder), or drug abuse will not be included as subjects. In addition, a score of 11 or greater on the Mini Mental Status Exam will be required to insure that subject can participate effectively in the study protocol. Because of potential effects on cognition and hemodynamic response, subjects currently taking benzodiazepines, narcotics, neuroleptics, anticonvulsants, antispasticity agents or psychostimulants will not be included.

In addition, any patient that is on medications that may interact with any of the study medications (e.g. birth control bills or cyclosporin). Psychiatric symptoms and substance abuse history will be obtained using a structured psychiatric interview, the Diagnostic Interview Schedule 129DIS. In addition patients with history of drug dependency, hypertension out of control, significant cardiac disease, or inability to undergo MRI. (e.g. metalworker, Medtronic infusion pump)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-08; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
mPASAT | Pre-Treatment, Post-Treatment
Dispersion of fMRI signal | Pre-Treatment, Post-Treatment
Simple Vigilance Task | Pre-Treatment, Post-Treatment
Neuropsychological Battery (Digit Vigilance Task, California Verbal Learning Test, Digit Span and Continuous Performance Task) | Pre-Treatment, Post-Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elie P Elovic, M.D., Principal Investigator — Kessler Medical Rehabilitation Research & Education Corporation
Locations (1):
- Kessler Medical Rehabilitation Research & Education Corporation, West Orange, New Jersey, United States

REFERENCES:
- [Background] Baddeley A. Working memory. Science. 1992 Jan 31;255(5044):556-9. doi: 10.1126/science.1736359.
- [Background] Levin HS, Gary HE Jr, Eisenberg HM, Ruff RM, Barth JT, Kreutzer J, High WM Jr, Portman S, Foulkes MA, Jane JA, et al. Neurobehavioral outcome 1 year after severe head injury. Experience of the Traumatic Coma Data Bank. J Neurosurg. 1990 Nov;73(5):699-709. doi: 10.3171/jns.1990.73.5.0699. PMID 2213159
- [Background] McDowell S, Whyte J, D'Esposito M. Working memory impairments in traumatic brain injury: evidence from a dual-task paradigm. Neuropsychologia. 1997 Oct;35(10):1341-53. doi: 10.1016/s0028-3932(97)00082-1. PMID 9347480
- [Background] Ponsford J, Kinsella G. Attentional deficits following closed-head injury. J Clin Exp Neuropsychol. 1992 Sep;14(5):822-38. doi: 10.1080/01688639208402865. PMID 1474148
- [Background] Stuss DT, Ely P, Hugenholtz H, Richard MT, LaRochelle S, Poirier CA, Bell I. Subtle neuropsychological deficits in patients with good recovery after closed head injury. Neurosurgery. 1985 Jul;17(1):41-7. doi: 10.1227/00006123-198507000-00007. PMID 4022286
- [Background] McAllister TW, Saykin AJ, Flashman LA, Sparling MB, Johnson SC, Guerin SJ, Mamourian AC, Weaver JB, Yanofsky N. Brain activation during working memory 1 month after mild traumatic brain injury: a functional MRI study. Neurology. 1999 Oct 12;53(6):1300-8. doi: 10.1212/wnl.53.6.1300. PMID 10522888
- [Background] Thurman DJ, Alverson C, Dunn KA, Guerrero J, Sniezek JE. Traumatic brain injury in the United States: A public health perspective. J Head Trauma Rehabil. 1999 Dec;14(6):602-15. doi: 10.1097/00001199-199912000-00009. PMID 10671706
- [Background] Schootman M, Fuortes LJ. Ambulatory care for traumatic brain injuries in the US, 1995-1997. Brain Inj. 2000 Apr;14(4):373-81. doi: 10.1080/026990500120664. PMID 10815845
- [Background] Guerrero JL, Thurman DJ, Sniezek JE. Emergency department visits associated with traumatic brain injury: United States, 1995-1996. Brain Inj. 2000 Feb;14(2):181-6. PMID 10695573
- [Background] Smith EE, Jonides J, Koeppe RA. Dissociating verbal and spatial working memory using PET. Cereb Cortex. 1996 Jan-Feb;6(1):11-20. doi: 10.1093/cercor/6.1.11. PMID 8670634